CLINICAL TRIAL: NCT03609983
Title: Diet, Physical Activity, and Weight Trends Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: UTK IRB-18-04488-XP
Record Dates: First submitted 2018-06-17; First posted 2018-08-01 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Self-Regulation
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Intervention Model Description: A 3x2 mixed factorial design will be used, with a between-subject factor will of self-weighing group (daily weighing; weekly weighing; and no weighing control group) and within-subject factor will of time (prior to self-weighing and feedback and during self-weighing and feedback).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily Weighing (Experimental): Participants will weigh themselves daily and receive feedback daily.
  Interventions: Other: Daily weighing with daily feedback on weight
- Weekly Weighing (Experimental): Participants will weigh themselves weekly and receive feedback weekly.
  Interventions: Other: Weekly weighing with weekly feedback on weight
- No Weighing (No Intervention): Participants will refrain from weighing themselves.

INTERVENTIONS:
Other: Daily weighing with daily feedback on weight — Participants will weigh themselves using a Yunmai SE Scale one time each day upon rising from bed beginning in one week, every day for four weeks. After 2 weights have been collected, participants will begin to receive daily feedback on their change in weight and suggestions to maintain energy balance. They will receive an email stating, "Your weight today is _______. Your weight has (increased/decreased) _____ pounds since yesterday." If their weight has increased, the email will include one example of how to decrease their energy balance by 150 calories. If participants' weight has decreased, the email will include one example of how to increase energy balance by 150 calories.
  Arms: Daily Weighing
Other: Weekly weighing with weekly feedback on weight — Participants will weigh themselves using a Yunmai SE Scale one time each week upon rising from bed beginning the following day for four weeks. After 2 weights have been collected, participants will begin to receive weekly feedback on their change in weight and suggestions to maintain energy balance. They will receive an email stating, "Your weight today is _______. Your weight has (increased/decreased) _____ pounds since last week." If their weight has increased, the email will include one example of how to decrease their energy balance by 150 calories. If participants' weight has decreased, the email will include one example of how to increase energy balance by 150 calories.
  Arms: Weekly Weighing

SUMMARY:
The purpose of this investigation is to is to examine if self-weighing with feedback, in which the feedback is matched to the timeframe of self-weighing, in the absence of a standard behavioral intervention assists with the self-regulation of energy balance behaviors among young adults. Participants will be randomized to one of three groups: 1) daily weighing; 2) weekly weighing; 3) no weighing for 4 weeks.

DETAILED DESCRIPTION:
All eligible participants will be scheduled for a baseline assessment at the Healthy Eating and Activity Laboratory (HEAL) that will last approximately 60 minutes. During this assessment, interested participants will sign the consent form. After signing the consent from, eligibility will be confirmed by taking height and weight measures and completing questionnaires assessing eating disorder risk and unhealthy weight control behaviors. Participants will also be given questionnaires assessing self-esteem and mood. Demographic information and contact information will be obtained. Next, eligible participants will be registered for the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) and provided instructions on how to complete 24-hour recalls using ASA24. Throughout the next week, participants will be randomly emailed on three days to complete three 24-hour recalls (1 weekend day, 2 weekdays). Participants will also be given a SenseWear Armband and provided instructions on how to use and care for the Armband. Participants will be instructed to wear the Armband for a minimum of 10 hours each day for the next week. At the conclusion of the session, participants will be scheduled to return to HEAL lab one week later.

This session one week later will last approximately 30 minutes. The investigator will confirm through ASA24 that the participant successfully completed three 24-hour recalls. To confirm that the participant successfully wore the Armband for at least 10 hours on the days the 24-hour recalls were completed, the investigator will download the Armband data using SenseWear software. After it has been confirmed that the participant completed these diet and physical activity measures, the participant will be randomized to the daily weighing group, weekly weighing group, or no weighing control group based on weight status. Participants in all groups will be provided with a handout containing general nutrition information about how to build a healthy eating pattern based on the 2015-2020 Dietary Guidelines for Americans.

Daily Weighing- Participants in the daily weighing group will be given a Yunmai SE Weight Scale and instructions for its use. Next, participants will be given instructions to download the Yunmai mobile app and create a user profile. Participants will be instructed to weigh themselves using the Yunmai SE Scale and app one time each day upon rising from bed (and before noon) after urination and in light clothing beginning in one week, every day for four weeks. Participants will be instructed to only weigh themselves using the scale provided during the duration of the study and to not allow others in their household use the scale. A reminder text and email will be sent to the participant to remind them to begin weighing on the assigned day. If on any day the participant has not weighed by 11am, the participant will receive an email and text reminder. After 2 weights have been collected, participants will begin to receive daily feedback on their change in weight and suggestions to maintain energy balance. They will receive an email between 12-1pm with this feedback stating, "Your weight today is _______. Your weight has (increased/decreased) _____ pounds since yesterday." If their weight has increased, the email will also contain a message stating, "If your goal is to maintain your weight, you may consider decreasing your energy balance by 150 calories" and will include one example of how to decrease their energy balance by 150 calories. If participants' weight has decreased, the participants will receive a message in addition to their feedback on change in weight stating, "If your goal is to maintain your weight, you may consider increasing your energy balance by 150 calories" and will include one example of how to increase energy balance by 150 calories.

Weekly Weighing- Participants in the weekly weighing intervention group will be given a Yunmai SE Weight Scale and instructions for its use. Next, participants will be given instructions to download the Yunmai mobile app and create a user profile. Participants will be instructed to weigh themselves using the Yunmai SE Scale and app one time each week upon rising from bed (and before noon) after urination in light clothing beginning the following day for four weeks. Participants will be instructed to only weigh themselves using the scale provided during the duration of the study and to not allow others in their household use the scale. If the participant has not weighed by 11am, the participant will receive an email and text reminder. After two weights have been collected, participants will begin to receive weekly feedback on their week and suggestions to maintain energy balance. Feedback and suggestions will be given as previously described above.

No Weighing Control- Participants in the non-weighing control group will be asked to refrain from weighing themselves for the next four weeks.

At the conclusion of the session, participants will be scheduled to return to HEAL lab three weeks later. This session three weeks later will last approximately 5 minutes. Participants will receive the Armband and be instructed to wear the Armband for a minimum of 10 hours each day during for the next week and reminded on how to complete 24-hour recalls using ASA24. Throughout the next week, participants will be randomly emailed on three days to complete three 24-hour recalls (1 weekend day, 2 weekdays). At the end of session, the participants will be scheduled to return to HEAL lab one week later. This session one week later will last approximately 60 minutes. Participants will be weighed and measured and be asked to complete follow-up questionnaires for eating attitudes, binge eating, unhealthy weight control behaviors, mood, and self-esteem. Participants will also be asked questions regarding their thoughts and feelings about self-regulation. Participants will also return the Armband and Yunmai SE Scale (intervention groups only) to the researcher. Handouts generated from ASA24 and SenseWear software that summarize the participant's dietary intake data from ASA24 and physical activity data from the Armband will be provided to the participants.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 29 years
* body mass index (BMI) 19.0-29.9 kg/m^2
* weight goal of maintaining current weight/preventing weight gain
* own and iPhone or Android phone to download the Yunmai app for the scale used for self-weighing
* daily access to a computer with internet to complete dietary assessments online through ASA24
* regularly wake up before 12pm (noon) on weekdays (Monday-Friday) and weekend days (Saturday-Sunday)
* present on campus for time period required to complete the study

Exclusion Criteria:

* self-reported previous or current diagnoses of an eating disorder, or at risk for an eating disorder defined as a score of ≥20 on EAT-26 and/or a score >27 on BES, and/or report of any extreme unhealthy weight control behaviors
* participating in a program that sets dietary or physical activity goals
* health condition that influences eating or physical activity or requires a therapeutic diet or physical activity restrictions
* allergy to metal making the participant unable to wear BodyMedia SenseWear Armband.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
24-hour Dietary Recall | Change in diet from Week 1 to Week 5
  Dietary intake data for 24-hour recalls will be collected using the Automated Self-Administered 24-Hour (ASA24), Dietary Assessment Tool, version 2016, developed by the National Cancer Institute, Bethesda, MD. Participants will be registered for ASA24 at the baseline appointment. Throughout the week following the baseline appointment, participants will be randomly emailed on three days to complete three 24-hour recalls (1 weekend day, 2 weekdays) through ASA24. Participants will be randomly emailed again on three days to complete three 24-hour recalls (1 weekend day, 2 weekdays) through ASA24 during the final week of the self-weighing condition.
Physical Activity | Change in physical activity from Week 1 to Week 5
  Activity will be collected with SenseWear Armbands worn by participants for at least 10 hours/day for one week after the baseline appointment and during the final week of the self-weighing condition. The SenseWear Armband utilizes a 2-axis accelerometer to detect motion, a heat flux sensor, galvanic skin response sensor (GSR), skin temperature sensor, and a near-body ambient temperature to calculate energy expenditure. The dependent variables will be total energy expenditure (kJ), moderate- to vigorous-intensity physical activity duration (3.0 METs and higher), and number of steps.

SECONDARY OUTCOMES:
Weight | Baseline appointment and follow-up appointment 5 weeks later
  Weight will be assessed by an electronic scale using standard procedures, with participants wearing light clothing, without shoes.
Eating Attitudes | Baseline appointment and follow-up appointment 5 weeks later
  The Eating Attitudes Test (EAT-26) will be administered to participants at baseline and follow-up assessments. This 26-item self-report questionnaire is designed to measure symptoms and concerns that are characteristic of eating disorders. A high score (≥20) indicates concerns regarding body weight, body shape, and eating.
Binge Eating | Baseline appointment and follow-up appointment 5 weeks later
  The Binge Eating Scale (BES) will be administered to participants at baseline and follow-up assessments. This 16-item self-report questionnaire is designed to capture the behavioral, cognitive, and emotional features of binge eating that may be indicative of an eating disorder. A high score (>27) indicates severe binge eating problems.
Unhealthy Weight-Control Behaviors | Baseline appointment and follow-up appointment 5 weeks later
  To assess the presence of extreme unhealthy weight control behaviors (UWCB), the following question will be asked to participants at baseline and follow-up assessments: 'Have you done any of the following things in order to lose weight or keep from gaining weight during the past 4 weeks? (yes or no for each method).' Behaviors categorized as less extreme UWCB will include (1) fasted, (2) ate very little food, (3) used a food substitute (e.g. Slim-fast), (4) skipped meals and (5) smoked more cigarettes; and behaviors categorized as extreme UWCB will include (6) took diet pills, (7) made yourself vomit, (8) used laxatives and (9) used diuretics.
Self-Esteem | Baseline appointment and follow-up appointment 5 weeks later
  Self-esteem will be assessed at baseline and follow-up using the State Self Esteem Scale (SSES).This is a 20-item scale that measures a participant's self-esteem at a given point in time. The 20 items are subdivided into 3 components of self-esteem: (1) performance self-esteem, social self- esteem, and appearance self-esteem. All items are answered using a 5-point scale (1= not at all, 2= a little bit, 3= somewhat, 4= very much, 5= extremely) with a higher score indicating greater self-esteem.
Mood | Baseline appointment and follow-up appointment 5 weeks later
  Mood will be assessed at baseline and follow-up using the Profile of Mood States (POMS).This is a 65-item questionnaire designed to evaluate individuals within seven different mood domains: fatigue-inertia, anger-hostility, vigor-activity, confusion- bewilderment, depression-dejection, tension-anxiety, and friendliness. The depression-dejection and tension-anxiety subscales will be used for this study. The tension-anxiety subscale includes 9 items with scores ranging from 0-36, and the depression-depression includes 15 items with scores ranging from 0-60. Items are answered using a 5-point scale (0= not at all, 1= a little bit, 2= somewhat, 3= very much, 4= extremely) with a higher score indicating higher levels of anxiety and/or depression.
Participant Feedback | End of study 5 weeks after baseline appointment
  At follow-up, participants in the weighing conditions will be asked their thoughts and feelings about self-regulation. This will be assessed with the following questions: 1) 1. What is your current weight goal? (maintain current weight, lose weight, gain weight); 2) If you saw your weight on the scale go up from the previous day/week, how did you respond?; 3) If you saw the number on the scale go down from the previous day/week, how did you respond?; 4) If you saw the number on the scale remain the same from the previous day/week, how did you respond?

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Prushinski, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. J Am Diet Assoc. 2011 Jan;111(1):92-102. doi: 10.1016/j.jada.2010.10.008. PMID 21185970
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] The National Cancer Institute. Automated Self-Administered 24-Hour Dietary Assessment Tool. The National Cancer Institute. https://epi.grants.cancer.gov/asa24/. Published 2016. Accessed January 18, 2018.
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Lopez-Guimera G, Neumark-Sztainer D, Hannan P, Fauquet J, Loth K, Sanchez-Carracedo D. Unhealthy weight-control behaviours, dieting and weight status: a cross-cultural comparison between North American and Spanish adolescents. Eur Eat Disord Rev. 2013 Jul;21(4):276-83. doi: 10.1002/erv.2206. Epub 2012 Oct 11. PMID 23055262
- [Background] Heatherton TF, Polivy J. Development and validation of a scale for measuring state self-esteem. Journal of Personality and Social Psychology. 1991;60(6):895.
- [Background] McNair D, Lorr M, Droppleman L. Profile of mood state manual. San Diego (CA): Educational and Industrial Testing Service. 1971.
- [Background] Garner DM. Eating attitudes test (EAT-26): Scoring and interpretation. http://www.eat-26.com/Docs/EAT-26IntpretScoring-Test-3-20-10.pdf. Accessed February 20, 2018.
- [Background] Cotter EW, Kelly NR. Binge Eating Scale (BES). In: Wade T, ed. Encyclopedia of Feeding and Eating Disorders. Singapore: Springer Singapore; 2016:1-5.
- [Background] Marcus MD, Wing RR, Hopkins J. Obese binge eaters: affect, cognitions, and response to behavioural weight control. J Consult Clin Psychol. 1988 Jun;56(3):433-9. doi: 10.1037//0022-006x.56.3.433. No abstract available. PMID 3397436